CLINICAL TRIAL: NCT05617781
Title: Analysis of Empathy in Patients With Post-traumatic Stress Disorder Followed at the Hospital of Nice: Case-control Study
Brief Title: Empathy in Post-traumatic Stress Disorder in Comparaison to a Control Population
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22-PP-19
Record Dates: First submitted 2022-11-03; First posted 2022-11-15 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Mental Disorder; Post-traumatic Stress Disorder; Empathy
MeSH Terms: conditions — Mental Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control
  Interventions: Behavioral: Questionnary
- Patient
  Interventions: Behavioral: Questionnary

INTERVENTIONS:
Behavioral: Questionnary — The primary outcome of this study is to analyze the post-traumatic stress disorder's repercussions on empathy by passing the Interpersonal Reactivity Index (IRI)

SUMMARY:
It has been shown in the literature that the symptoms of post-traumatic stress disorder influence the quality of life of patients, in particular through the cognitive alterations they can cause. Social cognition is also itself impacted. It refers to the perception, interpretation and processing of information relating to the social environment and relationships. It is affected by the symptomatology of PTSD both in terms of the response to emotional stimuli, the perception of self and others, and the quality of intimate relationships. These elements lead to reflection on the origin of these alterations, in particular the impact of PTSD on the patient's empathy capacity, defined as the recognition and understanding of the feelings and emotions of another individual. This parameter is also little studied in the literature, only a study dating from 2010 finds a correlation between PTSD and empathy. It is in this context that the realization of a new study studying the capacity for empathy of patients with PTSD in comparison with a control group with a larger and more representative population was envisaged. The primary outcome of this study is to analyze the post-traumatic stress disorder's repercussions on empathy by passing the Interpersonal Reactivity Index (IRI) on patients in comparison with a control group. The first hypothesis is a lower total score but a higher personal distress sub-score in the PTSD population. The secondary outcomes are to describe the cofactors that can influence empathy in association or not with post-traumatic stress disorder: sociodemographic data (age, sex, education level…), traumatic event type determined through the "Inventory of Traumatogenic Events", human intervention, duration and severity of the disorder (evaluated by the Impact of Events Scale) … The number of subjects required was calculated at 19 patients and 19 controls.

ELIGIBILITY:
Any patient or controls who score positively off the diagnostic criteria for comorbidities such as major depressive episode, generalized anxiety disorder, psychotic disorder and autism spectrum disorder are not included. These criteria will be assessed through the MINI diagnostic interview and the Autism Spectrum Quotient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients included will be followed at the Hospital of Nice for post-traumatic stress disorder diagnosed according to the DSM-V criteria. They are volunteers, adults, French speakers. The control population will be randomly selected (advertising, social networks…), adults and French speakers too, having no follow-up or current psychiatric treatment.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Interpersonal Reactivity Index (IRI) | 1 visit for inclusion
  The Interpersonal Reactivity Index is a validated self-questionnaire allowing the measurement of empathy from 28 items. For each item, five rating levels are proposed in the form of a Likert scale ranging from 0 ("does not describe me at all") to 4 ("describes me completely"). The IRI is divided into four subscales of seven items corresponding to conceptual adaptation (tendency to spontaneously adopt the point of view of others in daily life), fantasy (tendency to imagine oneself in fictitious situations) , empathic concern (tendency to experience feelings of sympathy and compassion in response to the distress of others) and personal distress (tendency to experience distress and discomfort in response to the distress of others.) The score of each subscale therefore varies from 0 to 28 and the total score of the IRI is between 0 and 112.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No